

Teaching Subdirectorate Research Coordination

| R | F | C | F | P | Т | Ю | N | D | Α | T | F |
|---|---|---|---|---|---|---|---|---|---|---|---|

PROVISIONAL REGISTRATION

DO NOT FILL

### **REGISTRATION OF THE INVESTIGATION PROTOCOL**

1. GENERAL DATA

1.1 TITLE OF THE PROJECT

1.2 START DATE

"Effect of intravenous iron repletion on renal function in patients with

iron deficiency and acute kidney injury, clinical trial"

**FINISH DATE** 

| Start August 2022, end | d December 2023 | |
|--------------------------------|-----------------|-----------------|
| <u>1.4 PRINCIPAL</u><br>NAME : | LAST NAME | Chávez |
| PATERNAL: | | Iniguez |
| MATERNAL: | | |
| (C)· | NAMES | Jonathan Samuel |
| (S):<br>SPECIALTY: Nep | hrology | |
| SERVICE: Nephr | ology | |
| 1.5 THESIS DIRI | ECTOR | |
| NAME :<br>PATERNAL: | LASTNAME | Chávez |
| MATERNAL: | | Iniguez |
| | NAMES | Jonathan Samuel |
| (S):<br>SPECIALTY: Nep | hrology | |
| SERVICE: Nephr | ology | |

Version 2.0, 29 June 2023 HOSPITAL No. 278 SHCP 44280 TEL. 3614-5501, 3614-7244 GUADALAJARA, JAL



Ron

LASTNAME

Teaching Subdirectorate Research Coordination

NAME:

1.6 CO-MANAGER

| PATERNAL: | | |
|---|---|---|
| | | Magaña |
| MATERNAL: | NAMES | Ana Lucia |
| (S): | | |
| SPECIALTY: Hematolo | | |
| SERVICE: Hematology | / | |
| 1.7 ADVISOR | | |
| NAME : | LAST NAME | |
| PATERNAL: | | |
| MATERNAL: | NAMEO | |
| (S): | NAMES | |
| SPECIALTY: | | |
| SERVICE: | | |
| 1.8 PARTICIPATING IN | STITUTIONS | |
| _ | | dalajara Fray Antonio Alcalde |
| INSTITUTION: | | dalajara i Tay Amomo Alcaide |
| AGREEMENT: | without agreement | |
| ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | |
| INSTITUTION: | | |
| AGREEMENT: | | |
| INSTITUTION: | | |
| A ODEENIEN'T | | |
| AGREEMENT: | Version 2.0 | 29 June 2023 |
| HOSPITAL No. 278 S | | 5501 3614-7244 GHADALA IARA TAL |



Teaching Subdirectorate Research Coordination

### 2.1 PROJECT SUMMARY

The purpose of this clinical trial is to carry out research on the effect on hemoglobin and renal function of the intravenous administration of iron dextran as a repletion strategy in patients with iron deficiency anemia and acute kidney injury, in which the patient You may benefit from this medication since it is expected to correct anemia, iron deficiency and renal function parameters, when compared with a control group (placebo), the safety of the drug will also be evaluated by recording adverse effects. I will point out with the patient the risks and benefits of including her in this type of study and I will answer all the doubts that arise, and I will also immediately report any serious adverse effect to the research ethics committee.



Teaching Subdirectorate Research Coordination

### 2.2 INTRODUCTION

Acute kidney damage is a complication that occurs in up to 30% of hospitalized patients. Iron deficiency has a high incidence in the population of critically ill patients and has been associated with multiple complications such as the development of anemia and renal dysfunction. The presence of iron deficiency, anemia and acute kidney injury is a common combination in critically ill patients and iron deficiency has been shown to promote mitochondrial dysfunction and this can be improved with intravenous iron correction, as has happened in clinical trials of patients with failure exacerbated cardiac arrest, improving its clinical evolution.

The kidney is the second organ with the most mitochondria and mitochondrial dysfunction is a new therapeutic goal in acute kidney injury. It is possible that this combination is associated with an unfavorable clinical course in these patients.

## 2.3 JUSTIFICATION

There is insufficient evidence for the implementation of intravenous iron in order to improve the parameters of iron deficiency anemia in patients with acute kidney injury.

To our knowledge, there is no clinical trial that has explored our objectives.

Version 2.0, 29 June 2023

Effect of intravenous iron repletion on renal function in patients with iron deficiency and acute kidney injury, clinical trial. June 2023, HCG/CEI-1232/22



Teaching Subdirectorate Research Coordination

### 2.4 SCIENTIFIC BACKGROUND

Acute kidney injury (ARD) is a serious complication that is independently associated with poor outcomes [1, 2]. Approximately one in five patients with non-severe sepsis develops AKI [3], which increases to two-thirds in critically ill patients. About 50% of ICU patients with AKI die (4-12), and those who survive an episode of AKI have a higher risk of progressing to chronic kidney disease (CKD). Currently, there are few pharmacological therapeutic options available to prevent or treat AKI, and management is limited to alleviating hemodynamic and toxic renal lesions. support measures, such as dialysis.

Iron deficiency occurs in up to 30% of hospitalized patients and has been linked to worse clinical evolution, even in the absence of anemia. This iron deficiency is worse even when anemia figures are reached. It has been documented that critically ill patients develop anemia as part of the process of their pathology. It has been seen that during processes of exacerbation of pathologies such as heart failure, the administration of intravenous iron avoids the probability of hospitalization and clinical evolution (13-16). It has been shown that in DRA there is mitochondrial dysfunction (17), specifically in the renal tubule where the greatest amount of mitochondria isconcentrated,


Effect of intravenous iron repletion on renal function in patients with iron deficiency and acute kidney injury, clinical trial. June 2023, HCG/CEI-1232/22



Teaching Subdirectorate Research Coordination

#### 2.5 OBJECTIVES

### Primary objective:

The endpoint of interest was the proportion of patients meeting one or more criteria for Major Adverse Kidney Events within 30 days (MAKE30): in-hospital mortality; receipt of new RRT; or persistent renal dysfunction.

In hospital mortality was defined as death from any cause prior to hospital discharge censored at 30 days after ICU admission. Receipt of new RRT was defined as receipt of any modality of RRT between ICU admission and the first of (1) hospital discharge or (2) 30 days in a patient not known to have received RRT prior to ICU admission. Persistent renal dysfunction was defined as a final serum creatinine value before hospital discharge (censored at 30 days after enrollment) that was  $\geq$  200 % of the baseline creatinine value.

And will be evaluated at 60 and 90 days.

**Secondary objectives**: all the following will be at hospital discharge and 28 days after hospital discharge between the intervention group (iron replacement) compared to the control group (placebo).

- ferritin value, (pg/dL)
- transferrin saturation (%)
- Hemoglobin (g/dL)
- serum creatinine (mg/dL)
- start of renal support therapy (any type of renal support such as: intermittent hemodialysis, peritoneal dialysis or continuous therapies)
- recovery of renal function, considered as a decrease in serum creatinine and approaching <0.3mg/dL of basal creatinine</li>
- death

## **Exploratory objectives:**

 safety of intravenous iron administration compared to placebo: assessed by the occurrence of adverse events such as allergic reaction, hypotension, dyspnea, rash, erythema. These will be evaluated during

HOSPITAL No. 278 SHCP 44280 TEL. 3614-5501, 3614-7244 GUADALAJARA, JAL



drug administration and during hospitalization frequently every 24 hours by the nephrology staff, including the study investigators.



Teaching Subdirectorate Research Coordination

#### 2.6 HYPOTHESIS

Our hypothesis is that intravenous iron dextran repletion during the treatment of acute kidney injury will improve renal function parameters, iron deficiency, anemia, and also that it will be safe compared to placebo.

### 2. DESIGN OF THE STUDY

Randomized placebo-controlled clinical trial, randomization method in blocks of 5 by frequency of occurrence. In patients with acute kidney injury, they will be randomized to receive the administration of intravenous iron dextran in a single exhibition according to the Mg provided by the Virizzi formula compared to placebo.

The sample size determined 55 patients per group, with a standard deviation of 1.5.

n = 
$$[(Z_{\alpha/2}+z_{\beta})_2 \times \{2(or)_2\}]/(\mu 1 - \mu 2)_2$$
  
n =  $[(1.96+0.84)_2 \times \{2(1.5)_2\}]/(10.8 - 10)_2$   
n=**55.125**

n = sample size required in each group  $\mu$ 1- $\mu$ 2 = clinically significant difference = 0.8 or = standard deviation = 1.5  $z_{\alpha/2}$ : 1.96  $z_{\beta}$ : 0.84


Effect of intravenous iron repletion on renal function in patients with iron deficiency and acute kidney injury, clinical trial. June 2023, HCG/CEI-1232/22



Teaching Subdirectorate Research Coordination

The randomization process by random assignment was carried out with the toolNCI Clinical Trial Randomization Tool:

https://ctrandomization.cancer.gov/

Sequences have been generated for each arm and stratum of your trial using maximum asymptotic randomization.

| group | Subject | Assignment | Assigned Arm Index |
|-------|---------|--------------|-----------------------------|
| all | 1 | placebo | 2 |
| all | 2 | Dextran Iron | 1 |
| all | 3 | Dextran Iron | 1 |
| all | 4 | placebo | 2 |
| all | 5 | Dextran Iron | 1 |
| all | 6 | placebo | 2 |
| all | 7 | placebo | 2 |
| all | 8 | Dextran Iron | 1 |
| all | 9 | placebo | 2 |
| all | 10 | Dextran Iron | 1 |
| all | 11 | Dextran Iron | 1 |
| all | 12 | placebo | 2 |
| all | 13 | Dextran Iron | 1 |
| all | 14 | Dextran Iron | 1 |
| all | | placebo | 2 |
| | 15 | | |
| all | 16 | Dextran Iron | 1 |
| all | 17 | Dextran Iron | 1 |
| all | 18 | placebo | 2 |
| all | 19 | placebo | 2 |
| all | 20 | Dextran Iron | 1 Varaian 2.0. 20 Juna 2022 |
| all | 21 | Dextran Iron | Version 2.0, 29 June 2023 |
| all | 22 | placebo | 2 |

HOSPITAL No. 278 SHCP 44280 TEL. 3614-5501, 3614-7244 GUADALAJARA, JAL



all

23

Dextran Iron

1



## Teaching Subdirectorate Research Coordination

| all | 24 | placebo | 2 |
|-----|----|--------------|-------------|
| all | 25 | placebo | 2 |
| all | 26 | placebo | 2 |
| all | 27 | Dextran Iron | 1 |
| all | 28 | placebo | 2 |
| all | 29 | placebo | 2 |
| all | 30 | Dextran Iron | 1 |
| all | 31 | placebo | 2 |
| all | 32 | Dextran Iron | 1 |
| all | 33 | placebo | 2 |
| all | 34 | placebo | 2 |
| all | 35 | placebo | 2 |
| all | 36 | Dextran Iron | 1 |
| all | 37 | Dextran Iron | 1 |
| all | 38 | Dextran Iron | 1 |
| all | 39 | Dextran Iron | 1 |
| all | 40 | Dextran Iron | 1 |
| all | 41 | placebo | 2 |
| all | 42 | placebo | 2 |
| all | 43 | Dextran Iron | 1 |
| all | 44 | placebo | 2 |
| all | 45 | placebo | 2 |
| all | 46 | Dextran Iron | 1 |
| all | 47 | Dextran Iron | 1 |
| all | 48 | placebo | 2 |
| all | 49 | Dextran Iron | 1 |
| all | 50 | placebo | 2 |
| all | 51 | placebo | 2 |
| all | 52 | Dextran Iron | 1 |
| all | 53 | placebo | 2 |
| all | 54 | placebo | |
| all | 55 | Dextran Iron | 2<br>1<br>2 |
| all | 56 | placebo | 2 |
| all | 57 | Dextran Iron | 1 |
| all | 58 | Dextran Iron | 1 |


HOSPITAL No. 278 SHCP 44280 TEL. 3614-5501, 3614-7244 GUADALAJARA, JAL



## Teaching Subdirectorate Research Coordination

| all | 59 | Dextran Iron | 1 |
|-----|----|--------------|---------------------------------|
| all | 60 | Dextran Iron | 1 |
| all | 61 | placebo | 2 |
| all | 62 | placebo | 2 |
| all | 63 | Dextran Iron | 1 |
| all | 64 | placebo | 2 |
| all | 65 | Dextran Iron | 1 |
| all | 66 | Dextran Iron | 1 |
| all | 67 | placebo | 2 |
| all | 68 | placebo | 2 |
| all | 69 | placebo | 2 |
| all | 70 | placebo | 1<br>2<br>2<br>2<br>2<br>2<br>2 |
| all | 71 | placebo | 2 |
| all | 72 | Dextran Iron | 1 |
| all | 73 | Dextran Iron | 1 |
| all | 74 | Dextran Iron | 1 |
| all | 75 | Dextran Iron | 1 |
| all | 76 | placebo | 2 |
| all | 77 | placebo | 2<br>2<br>2<br>1 |
| all | 78 | placebo | 2 |
| all | 79 | Dextran Iron | |
| all | 80 | Dextran Iron | 1 |
| all | 81 | placebo | 2 |
| all | 82 | Dextran Iron | 1 |
| all | 83 | Dextran Iron | 1 |
| all | 84 | placebo | 2 |
| all | 85 | Dextran Iron | 1 |
| all | 86 | placebo | 2 |
| all | 87 | Dextran Iron | 1 |
| all | 88 | placebo | 2 |
| all | 89 | Dextran Iron | 1 |
| all | 90 | Dextran Iron | 1 |
| all | 91 | placebo | |
| all | 92 | Dextran Iron | 2<br>1<br>2 |
| all | 93 | placebo | 2 |




## Teaching Subdirectorate Research Coordination

| all | 94 | placebo | 2 | |
|-----|-----|--------------|---|---------------------------|
| all | 95 | placebo | 2 | |
| all | 96 | placebo | 2 | |
| all | 97 | placebo | 2 | |
| all | 98 | Dextran Iron | 1 | |
| all | 99 | Dextran Iron | 1 | |
| all | 100 | placebo | 2 | |
| all | 101 | Dextran Iron | 1 | |
| all | 102 | placebo | 2 | |
| all | 103 | Dextran Iron | 1 | |
| all | 104 | Dextran Iron | 1 | |
| all | 105 | placebo | 2 | |
| all | 106 | placebo | 2 | |
| all | 107 | placebo | 2 | |
| all | 108 | Dextran Iron | 1 | |
| all | 109 | placebo | 2 | |
| all | 110 | Dextran Iron | 1 | |
| all | 111 | Dextran Iron | 1 | |
| all | 112 | placebo | 2 | |
| all | 113 | Dextran Iron | 1 | |
| all | 114 | Dextran Iron | 1 | |
| all | 115 | placebo | 2 | |
| all | 116 | placebo | 2 | |
| all | 117 | Dextran Iron | 1 | |
| all | 118 | Dextran Iron | 1 | |
| all | 119 | placebo | 2 | Version 2.0, 29 June 2023 |
| all | 120 | placebo | 2 | |

, and members of the nephrology staff, blinded to the allocation groups, administered the drugs to each patient every day.

All patients will have a detailed medical history and physical examination. Complete blood count, serum creatinine, serum urea, serum urea nitrogen, serum electrolytes, and blood test parameters were measured daily.



Teaching Subdirectorate Research Coordination

urine. The test will be presented in accordance with the CONSORT 2010 explanation and elaboration guide. Continuous variables will be presented as mean (SD) when they are normally distributed or as medians (interquartile range [IQR]) in the case of abnormal distribution, following the test Shapiro-Wilk. One way ANOVA was used to compare differences between groups. Categorical variables expressed as proportions will be compared with Fisher's x2 test or the exact test, as appropriate. For the rest of the tests, p values were two-tailed; p <0.05 will be considered statistically significant. Statistical analysis and graphics will be performed with the statistical software MedCalc (Ostend, Belgium, see 19.1.3).

## 4.1 INCLUSION AND EXCLUSION CRITERIA

### criteria of inclusion:

Hospitalized patients with ARD, will be defined as the diagnosis using the KDIGO criteria of serum creatinine (Cr); Patients with AKI > 18 and <85 years, baseline creatinine <2 mg/dL and with written informed consent will be included.

Iron deficiency according to the criteria of the 2: serum iron <13 ng/dL, transferrin saturation <20%.



Teaching Subdirectorate Research Coordination

### 4.2 VARIABLES UNDER STUDY

Exposure variable is the administration of iron dextran in an infusion bolus as a loading strategy.

Dependent variables will be the value of renal function by eGFR, hemoglobin, iron deficiency, renal function and safety parameters.

### 4.4 ETHICAL ASPECTS

YO. RESEARCH WITHOUT RISK RESEARCH WITH

II. MINIMAL RISK RESEARCH WITH RISK

XXXX

III. GREATER THAN MINIMAL

ANNEX LETTER OF CONSENT



Teaching Subdirectorate Research Coordination

## Letter of consent attached to the protocol

## Visual summary of the study





Teaching Subdirectorate Research Coordination

5.1 SCHEDULE OF ACTIVITIES ATTACH FORMAT



| Year<br>Teaching direction | 2 | | | | | | | | | | 2 | | | | | | | 2 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Research dination | 0 | | | | | | | | | | 0 | | | | | | | 0 | ı |
| | 2 | | | | | | | | | | 2 | | | | | | | 2 | |
| | 3 | | | | | | | | | | 2 | | | | | | | 4 | ı |
| | m | T | m | J | J | TO | S | ЕІТН | кN | .D | Al | ΝĐ | Τ | s | ЕПН | ₽Ν | οD. | A١ | ŧ |
| Month | to | В. | T | þοι | ko | RG. | Α | D. | EITH | гYс | Ν | οAI | ND. | Al | ND. | EITH | ⊪Yc | No | Į |
| | r | R. | A | ND | οL | EITHER | Р | yc | uV | C. | Al | NΒ. | EITH | ₽P | yc | υV | C. | A١ | ŀ |
| Definition of the | | | | | | | | | | | | | | | | | | | ı |
| question of | | | | | | | | | | | | | | | | | | | ı |
| investigation | | | | | | | | | | | | | | | | | | | l |
| construction of | | | | | | | | | | | | | | | | | | | ı |
| approach of | | | | | | | | | | | | | | | | | | | ı |
| problem | | | | | | | | | | | | | | | | | | | l |
| | | | | | | | | | | | | | | | | | | | Ì |
| population selection | | | | | | | | | | | | | | | | | | | ı |
| study | | | | | | | | | | | | | | | | | | | ı |
| | | | | | | | | | | | | | | | | | | | I |
| Database creation | | | | | | | | | | | | | | | | | | | |
| | | | | | | | | | | | | | | | | | | | l |
| | | | | | | | | | | | | | | | | | | | l |
| | | | | | | | | | | | | | | | | | | | I |
| data collection | | | | | | | | | | | | | | | | | | | |
| data ordering | | | | | | | | | | | | | | | | | | | |
| data ordering | | | | | | | | | | | | | | | | | | | ĺ |


Effect of intravenous iron repletion on renal function in patients with iron deficiency and acute kidney injury, clinical trial. June 2023, HCG/CEI-1232/22



Teaching Subdirectorate Research Coordination

| Analysis of data |
|---------------------------------------|
| Comparison with theoretical referents |
| Final report of the investigation |



Teaching Subdirectorate Research Coordination

### **DOCUMENTARY REFERENCES**

- 1. Lameire NH, Bagga A, Cruz D, De Maeseneer J, Endre Z, Kellum JA, Liu KD, Mehta RL, Pannu N, Van Biesen W, et al. Acute kidney injury: an increasing global concern. Lancet. 2013;382(9887):170–9.
- 2. Siew ED, Davenport A. The growth of acute kidney injury: a rising tide or just closer attention to detail? Kidney Int. 2015;87(1):46–61.
- 3. Murugan R, Karajala-Subramanyam V, Lee M, Yende S, Kong L, Carter M, Angus DC, Kellum JA. Acute kidney injury in non-severe pneumonia is associated with an increased immune response and lower survival. Kidney Int. 2010;77(6):527–35.
- 4. Nisula S, Kaukonen KM, Vaara ST, Korhonen AM, Poukkanen M, Karlsson S, Haapio M, Inkinen O, Parviainen I, Suojaranta-Ylinen R, et al. Incidence, risk factors and 90-day mortality of patients with acute kidney injury in Finnish intensive care units: the FINNAKI study. Intensive Care Med. 2013;39(3):420–8.
- 5. Bagshaw SM, George C, Dinu I, Bellomo R. A multi-centre evaluation of the RIFLE criteria for early acute kidney injury in critically ill patients. Nephrol Dial Transplant. 2008;23(4):1203–10.
- 6. Ostermann M, Chang RW. Acute kidney injury in the intensive care unit according to RIFLE. Crit Care Med. 2007;35(8):1837–43. quiz 1852
- 7. Hoste EA, Clermont G, Kersten A, Venkataraman R, Angus DC, De Bacquer D, Kellum JA: RIFLE criteria for acute kidney injury are associated with hospital mortality in critically ill patients: a cohort analysis. CritCare 2006, 10(3):R73.
- 8. Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, et al. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015;41(8):1411–23.




## Teaching Subdirectorate Research Coordination

- 9. Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D, et al. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006;34(2):344–53.
- 10. Case J, Khan S, Khalid R, Khan A. Epidemiology of acute kidney injury in the intensive care unit. Crit Care Res Pract. 2013;2013:479730.
- 11. Chawla LS, Amdur RL, Amodeo S, Kimmel PL, Palant CE. The severity of acute kidney injury predicts progression to chronic kidney disease. Kidney Int. 2011;79(12):1361–9.
- 12. Wang HE, Muntner P, Chertow GM, Warnock DG. Acute kidney injury and mortality in hospitalized patients. Am J Nephrol. 2012;35(4):349-55.
- 13. Zarjou A, Agarwal A. Sepsis and acute kidney injury. J Am Soc Nephrol. 2011;22(6):999–1006.
- 14.- Andreini C, Putignano V, Rosato A, Banci L. The human iron-proteome. Metallomics. 2018 Sep 19;10(9):1223-1231. doi: 10.1039/c8mt00146d. PMID: 30095136.
- 15.-Alnuwaysir RIS, Hoes MF, van Veldhuisen DJ, van der Meer P, Beverborg NG. Iron deficiency in heart failure: mechanisms and pathophysiology. J Clin Med. 2021 Dec 27;11(1):125. doi: 10.3390/jcm11010125. PMID: 35011874; PMCID: PMC8745653.
- 16.- Melenovsky V, Petrak J, Mracek T, Benes J, Borlaug BA, Nuskova H, Pluhacek T, Spatenka J, Kovalcikova J, Drahota Z, Kautzner J, Pirk J, Houstek J. Myocardial iron content and mitochondrial function in human Heart failure: a direct tissue analysis. Eur J Heart Fail. 2017 Apr;19(4):522-530. doi: 10.1002/ejhf.640. Epub 2016 Sep 19. PMID: 27647766.




Teaching Subdirectorate Research Coordination

17. Hepokoski M, Singh P. Mitochondria as mediators of systemic inflammation and organ cross talk in acute kidney injury. Am J Physiol Renal Physiol. 2022 Jun 1;322(6):F589-F596. doi: 10.1152/ajprenal.00372.2021. Epub 2022 Apr 4. PMID: 35379000; PMCID: PMC9054254.